CLINICAL TRIAL: NCT00265811
Title: Adjuvant Treatment of Fully Resected Stage III Colon Cancer With FOLFOX-4 Versus FOLFOX-4 Plus Cetuximab
Brief Title: Combination Chemotherapy With or Without Cetuximab in Treating Patients With Stage III Colon Cancer That Was Completely Removed By Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000453839; FFCD-PETACC-8 (Other: FFCD); EU-20547; 2005-003463-23 (EudraCT Number); PETACC-8; MERCK-FFCD-PETACC-8
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; adenocarcinoma of the colon
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Folfox protocol; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Folfox+Cetuximab (Experimental): FOLFOX-4 Cetuximab alone every 2 weeks
  Interventions: Drug: Folfox; Drug: Cetuximab
- Folfox (Active Comparator): FOLFOX-4 alone every 2 weeks
  Interventions: Drug: Folfox

INTERVENTIONS:
Drug: Folfox
Drug: Cetuximab
  Arms: Folfox+Cetuximab

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, leucovorin, or fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Cetuximab may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving combination chemotherapy with or without cetuximab after surgery may kill any remaining tumor cells and keep colon cancer from coming back. It is not yet known whether giving combination chemotherapy together with cetuximab is more effective than giving combination chemotherapy alone in treating colon cancer.

PURPOSE: This randomized phase III trial is studying combination chemotherapy and cetuximab to see how well they work compared to combination chemotherapy alone in treating patients with stage III colon cancer that was completely removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the disease-free survival rates in patients with completely resected stage III colon cancer treated with adjuvant oxaliplatin, leucovorin calcium, and fluorouracil with vs without cetuximab.

Secondary

* Compare the 3-year disease-free survival rate and 5-year overall survival rate in patients treated with these regimens.
* Compare the overall survival of patients treated with these regimens.
* Compare the treatment compliance of patients treated with these regimens.
* Determine the prognostic factors and markers predictive for relapse and/or treatment efficacy in patients treated with these regimens.
* Compare the safety of these regimens in these patients.

OUTLINE: This is an open-label, randomized, controlled, multicenter study. Patients are stratified according to obstruction/perforation status (no obstruction and no perforation vs obstruction and/or perforation), N stage (N1 vs N2), and T stage (T1-3 vs T4). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oxaliplatin IV over 2 hours on day 1 and leucovorin calcium IV over 2 hours and fluorouracil IV continuously over 22 hours on days 1 and 2.
* Arm II: Patients receive chemotherapy as in arm I plus cetuximab IV over 1-2 hours on days 1 and 8.

In both arms, treatment repeats every 14 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for approximately 5 years.

PROJECTED ACCRUAL: A total of 2,000 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage III adenocarcinoma of the colon
* Must have undergone curative resection (R0) within the past 28-56 days

  * No radiotherapy prior to surgery
* carcinoembryonic antigen (CEA) ≤ 1.5 times upper limit of normal (ULN) after surgery
* No rectal cancer located within 15 cm from the anal verge by endoscopy or under the peritoneal reflection at surgery
* No metastatic spread at baseline assessment
* No prior or concurrent CNS disease by physical exam

PATIENT CHARACTERISTICS:

Performance status

* WHO 0-1

Life expectancy

* At least 5 years

Hematopoietic

* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL

Hepatic

* Bilirubin ≤ 1.5 times ULN
* AST and ALT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 1.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No coronary artery disease
* No myocardial infarction within the past 12 months
* No high risk of uncontrolled arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No inflammatory bowel disease
* No other malignancy within the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix
* No significant traumatic injury within the past 28 days
* No known hypersensitivity to any of the components of the study drugs
* No medical, geographical, sociological, psychological, or legal condition that would preclude study participation
* No peripheral neuropathy ≥ grade 1
* No other significant disease that would preclude study participation

PRIOR CONCURRENT THERAPY:

Chemotherapy

* No prior chemotherapy

Radiotherapy

* See Disease Characteristics
* No prior abdominal or pelvic irradiation

Surgery

* See Disease Characteristics
* Recovered from prior surgery
* More than 28 days since prior major surgical procedure or open biopsy
* No concurrent major surgical procedure

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2559 (Actual)
Dates: Start 2005-11 (Actual); Primary Completion 2009-11 (Actual); Study Completion 2010-06-22 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 3-years DFS
  DFS time in the ITT KRAS wild-type population

SECONDARY OUTCOMES:
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Julien Taieb, MD, Study Chair — CHU Pitie-Salpetriere
Locations (8):
- France (8):
  - Hopital Duffaut, Avignon
  - CHU de Caen, Caen
  - Hopital Robert Boulin, Libourne
  - Hopital Bichat - Claude Bernard, Paris
  - CHU Pitie-Salpetriere, Paris
  - Hopital Tenon, Paris
  - Centre Hospitalier Yves Le Foll, Saint-Brieuc
  - Nouvelle Clinique Generale, Valence

REFERENCES:
- [Result] Taieb J, Puig PL, Bedenne L. Cetuximab plus FOLFOX-4 for fully resected stage III colon carcinoma: scientific background and the ongoing PETACC-8 trial. Expert Rev Anticancer Ther. 2008 Feb;8(2):183-9. doi: 10.1586/14737140.8.2.183. PMID 18279058
- [Result] Taieb J, Tabernero J, Mini E, Subtil F, Folprecht G, Van Laethem JL, Thaler J, Bridgewater J, Petersen LN, Blons H, Collette L, Van Cutsem E, Rougier P, Salazar R, Bedenne L, Emile JF, Laurent-Puig P, Lepage C; PETACC-8 Study Investigators. Oxaliplatin, fluorouracil, and leucovorin with or without cetuximab in patients with resected stage III colon cancer (PETACC-8): an open-label, randomised phase 3 trial. Lancet Oncol. 2014 Jul;15(8):862-73. doi: 10.1016/S1470-2045(14)70227-X. Epub 2014 Jun 11. PMID 24928083
- [Derived] Gallois C, Shi Q, Meyers JP, Iveson T, Alberts SR, de Gramont A, Sobrero AF, Haller DG, Oki E, Shields AF, Goldberg RM, Kerr R, Lonardi S, Yothers G, Kelly C, Boukovinas I, Labianca R, Sinicrope FA, Souglakos I, Yoshino T, Meyerhardt JA, Andre T, Papamichael D, Taieb J. Prognostic Impact of Early Treatment and Oxaliplatin Discontinuation in Patients With Stage III Colon Cancer: An ACCENT/IDEA Pooled Analysis of 11 Adjuvant Trials. J Clin Oncol. 2023 Feb 1;41(4):803-815. doi: 10.1200/JCO.21.02726. Epub 2022 Oct 28. PMID 36306483
- [Derived] Cohen R, Taieb J, Fiskum J, Yothers G, Goldberg R, Yoshino T, Alberts S, Allegra C, de Gramont A, Seitz JF, O'Connell M, Haller D, Wolmark N, Erlichman C, Zaniboni A, Lonardi S, Kerr R, Grothey A, Sinicrope FA, Andre T, Shi Q. Microsatellite Instability in Patients With Stage III Colon Cancer Receiving Fluoropyrimidine With or Without Oxaliplatin: An ACCENT Pooled Analysis of 12 Adjuvant Trials. J Clin Oncol. 2021 Feb 20;39(6):642-651. doi: 10.1200/JCO.20.01600. Epub 2020 Dec 23. PMID 33356421
- [Derived] Salem ME, Yin J, Goldberg RM, Pederson LD, Wolmark N, Alberts SR, Taieb J, Marshall JL, Lonardi S, Yoshino T, Kerr RS, Yothers G, Grothey A, Andre T, De Gramont A, Shi Q. Evaluation of the change of outcomes over a 10-year period in patients with stage III colon cancer: pooled analysis of 6501 patients treated with fluorouracil, leucovorin, and oxaliplatin in the ACCENT database. Ann Oncol. 2020 Apr;31(4):480-486. doi: 10.1016/j.annonc.2019.12.007. Epub 2020 Jan 16. PMID 32085892
- [Derived] Taieb J, Shi Q, Pederson L, Alberts S, Wolmark N, Van Cutsem E, de Gramont A, Kerr R, Grothey A, Lonardi S, Yoshino T, Yothers G, Sinicrope FA, Zaanan A, Andre T. Prognosis of microsatellite instability and/or mismatch repair deficiency stage III colon cancer patients after disease recurrence following adjuvant treatment: results of an ACCENT pooled analysis of seven studies. Ann Oncol. 2019 Sep 1;30(9):1466-1471. doi: 10.1093/annonc/mdz208. PMID 31268130